CLINICAL TRIAL: NCT01880970
Title: Effect of Starter Formula With Synbiotics on Prevention of Gastro-intestinal Infections and All Infections With Fever in Full Term Infants
Brief Title: Effect of Starter Formula on Infection Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07.20.INF
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2014-07

CONDITIONS: Gastro-intestinal Infections; Infections With Fever
MeSH Terms: interventions — Proline; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Starter infant formula with pro and prebiotics (Active Comparator): starter infant formula from enrollment till 6 months of age, followed by a commercially available Nestlé follow-up formula from 6 to 12 months of age
  Interventions: Other: starter infant formula with pro and prebiotics
- starter infant formula without pro and prebiotics (Placebo Comparator): starter infant formula from enrollment till 6 months of age, followed by a commercially available Nestlé follow-up formula from 6 to 12 months of age
  Interventions: Other: Placebo comparator
- Breastfeeding group (No Intervention): exclusively breastfeeding during the first 3 months of age, followed by a commercially available Nestlé starter infant formula from 4 to 6 months of age (if applicable) and the follow-up infant formula from 6 to 12 months of age

INTERVENTIONS:
Other: starter infant formula with pro and prebiotics
  Arms: Starter infant formula with pro and prebiotics
Other: Placebo comparator
  Arms: starter infant formula without pro and prebiotics

SUMMARY:
The aim of this trial is to test the efficacy of an infant formula containing synbiotics on the prevention of gastro-intestinal infections.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infant
* Full term infant (≥ 37 weeks gestation; ≤ 42 weeks gestation)
* Age of infant is ≤ 13 days at the time of enrollment
* Birth weight ≥ 2500g and ≤ 4500g
* For the FF groups: The infant's mother has elected not to breastfeed
* For the BF group: The infant's mother has elected to fully breastfeed her baby, from enrollment to at least 3 months of age
* Having obtained his/her legal representative's informed consent

Exclusion Criteria:

* Congenital illness or malformation that may affect normal growth (especially immunodeficiencies)
* Significant pre-natal and/or post-natal diseases
* Perinatal antibiotic or infants on antibiotics at the time of inclusion
* Infants whose mother has had an acute infection during the last month of pregnancy
* Re-hospitalisation for more than 2 days in the first 14 days of life (exceptionally, infants re-hospitalized because of jaundice may be enrolled in the study)
* Receiving infant formula containing probiotics and/or prebiotics at the time of enrollment
* Newborn whose parents / caregivers cannot be expected to comply with treatment
* Newborn currently participating in another interventional clinical trial

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 477 (Actual)
Dates: Start 2008-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Diarrhea and all infections with fever | over 6 months and 1 year
  Mean event rate of diarrhea and all infections with fever per child over 6 months and 1 year

SECONDARY OUTCOMES:
Morbidity | over 6 months and 1 year
  Frequency of episodes of morbidity (adverse events), especially mean event rate of respiratory illnesses per child over 6 months and 1 year
Anthropometry | until 1 year
  Anthropometry (weight (kg), length (cm), head circumference (cm) and skin fold)
Digestive tolerance | until 1 year
  Digestive tolerance (stool characteristics and frequency, vomiting, regurgitation, frequency of colic)
Stool characteristics | at 3 and 6 months
  * Stool bacterial populations (Bifidobacteria, Lactobacilli Species, Clostridium, Bacteroides, Staphylococci epidermitis, presence or absence of B. lactis)
  * Stool pH
  * Stool and saliva S.IgA
  * Stool Alpha 1-antitrypsine as infection/inflammation marker

CONTACTS AND LOCATIONS:
Overall Officials: Jean Michel Hascoet, Prof., Principal Investigator — Maternité régionale de Nancy
Locations (7):
- France (3):
  - Hôpital de la Croix Rousse, Service de réanimation néonatale, Lyon
  - Hôpital Arnaud de Villeneuve, Service de pédiatrie 2, Montpellier
  - Maternité régionale de Nancy, Service de Néonatologie, Nancy
- Germany (3):
  - Charité Campus Virchow-Klinikum, Klinik für Geburtsmedizin, Berlin
  - Universitätsklinikum Gießen und Marburg, Zentrum für Kinderheilkunde und Jugendmedizin, Giessen
  - Klinikum Ernest von Bergmann, Klinik für Kinder- und Jugendmedizin, Potsdam
- Vrije Universiteit Medisch Centrum, Afdeling Kindergeneeskunde, Amsterdam, Netherlands